CLINICAL TRIAL: NCT05770817
Title: Surface-Knit and Reformulate CADENCE-Kids for Translation: The SKyRoCKeT Study
Brief Title: The SKyRoCKeT Study
Acronym: SKyRoCKeT
Status: Recruiting | Type: Observational
Sponsor: University of North Carolina, Charlotte (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Laura H Gunn, Principal Investigator, University of North Carolina, Charlotte
Other Study IDs: IRBIS-21-0460; 1R01HD105768-01A1 (NIH); 2021-1200 (Other Grant/Funding Number: University of North Carolina at Charlotte internal InfoEd grants management system record number)
Record Dates: First submitted 2023-03-01; First posted 2023-03-15 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Healthy
Keywords: cadence; steps; physical activity; physical activity intensity; metabolic equivalents (METs); cardiorespiratory fitness; indirect calorimetry; youth
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 6-20-year-old youth: 6-20-year-old youth
  Interventions: Other: N/A: SKyRoCKeT is an observational study

INTERVENTIONS:
Other: N/A: SKyRoCKeT is an observational study — None; this is an observational study

SUMMARY:
The SKyRoCKeT Study (Surface-Knit and Reformulate CADENCE-Kids for Translation) will recruit a sex- and age-balanced sample of 360 young people 6-20 years of age to develop an integrative, physiologically-coherent age-cadence-log(metabolic equivalent, MET) surface-based model, reformulate the prior R21 CADENCE-Kids study (1; NCT01989104) by providing individualized, more precise, age-specific and coherent cadence-intensity thresholds, investigate additional differences by anthropometric factors, and translate cadence-intensity thresholds to over-ground walking. The SKyRoCKeT Study is an innovative critical step to provide a coherent, interpretable, objectively monitored step-based intensity metric to inform (inter)national physical activity (PA) guidelines by transforming currently vague guidelines of PA intensity into quantifiable PA recommendations that can be of widespread use, which clinicians, young people, parents, and researchers can integrate into preventive care management and action plans for personalized care. The SKyRoCKeT Study will allow for a user-friendly, interpretable metric to more accurately inform public health/behavioral interventions, assessments, analyses, school-based health and physical education curricula and programs, and public health messages for young people and their caregivers.

DETAILED DESCRIPTION:
Specific Aims: The SKyRoCKeT Study will:

1. Expand CADENCE-Kids (1; NCT01989104) to innovatively surface-'knit' the age dimension through a continuous, unbiased-by-age, and physiologically-coherent age-cadence-log(MET) flexible surface approach without artificially-generated jumps between age ranges and with enhanced precision of cadence-intensity threshold estimates. This single surface will coherently transition between ages, borrow inter-age information, and be data-driven.
2. Reformulate CADENCE-Kids (1; NCT01989104) by providing age-specific cadence-intensity thresholds, calculated with enhanced precision for moderate and vigorous PA. Data will be objectively collected using a similar treadmill protocol to the R21-funded pilot study, with incrementally faster paces. Age-specific results will be compared to the pilot's age-range thresholds. A full running bout will now also be included. The investigators will concurrently collect cadence with direct observation and with multiple contemporary wearable technologies. Collecting cardiorespiratory fitness (CRF) and habitual PA data, the investigators will develop additional, innovative algorithms to predict relative intensity defined by lab-based indicators of oxygen uptake (%VO2peak, %VO2R), heart rate (%HRR, %HRmax), and rate of perceived of exertion (RPE) to facilitate computation of individually calibrated thresholds applicable to the free-living or habitual PA living condition. Investigators will assess differences in surfaces and cadence-intensity thresholds by sex and body mass index standard deviation scores (BMI SDS). Height- and/or leg-length-specific (hyper)surfaces will be explored as more precise alternatives to age.
3. Propel science forward innovatively through translation to over-ground walking. The investigators hypothesize that treadmill-set cadence-intensity thresholds will reliably translate and be useful for eliciting predictable metabolic costs during over-ground walking emblematic of free-living ambulatory behaviors.

Protocol/Procedures: 3 visits to the lab and 1 at home, free-living protocol

Screening: Screening questions will be completed online by potential participants (or their parents, where appropriate) and will take approximately 5 minutes. Following the initial recruitment web screener, potential participants (or their parents, where appropriate) will complete a telephone screener to confirm their responses. Potential participants (or their parents, where appropriate) will then attend a virtual or in-person orientation during which the study design procedures will be described in detail. Eligible potential participants who remain interested in the study will be scheduled for their first lab visit (with their parent/guardian if between 6-17 years of age).

Days of Testing in the Lab: Upon signing informed consent(s), participants must be fasted (no food for 4 hours before visit). Study procedures involving participants will be completed at the University of North Carolina at Charlotte. Visits 1 and 2 will be conducted at the Health Risk Assessment Laboratory (HRAL), and visit 3 will be conducted on an indoor track. Visit 1 will occur first and will be immediately followed by a week of free-living physical activity monitoring at home. Visit 2 will be completed once free-living, at-home monitoring is complete, and will be followed by visit 3.

Visit 1

* Demographic characteristic questions (approximately 5 minutes):

  o Participants will self-report their sex, race/ethnicity, and date of birth. Date of birth will be confirmed using a government issued ID (e.g. passport, driver's license or birth certificate).
* Anthropometrics (approximately 10 minutes):

  * Standing and seated height will be measured using a stadiometer.
  * Weight, BMI, and body fat percentage will be measured using a specialized scale; both weight with and without wearable devices will be measured.
* Instrument attachment, treadmill walking, free-living activities (approximately 140 minutes)

  * Participants will be fitted with multiple wearable devices (e.g., Fitbit, Apple Watch) to measure/monitor physical activity throughout the testing session.
  * Participants will then complete several low intensity free-living activities while their physical activity and oxygen uptake are concurrently measured. Specifically, participants will rest in a chair, watch a portion of a child-friendly movie while seated, and color in a coloring book while seated in a chair. Each activity will last for 5 minutes, and a 2-minute rest will occur between each activity
  * Participants will then begin the submaximal test by completing a series of walking bouts on a treadmill while their physical activity and oxygen uptake are concurrently measured. The walking bouts start at 0.5 miles per hour at a 0% incline and end at 6 miles per hour (0.5 miles per hour increments). A 2-minute rest will occur between each treadmill bout.
  * Following a 5-minute break, participants will then complete three additional free-living activities where physical activity and oxygen uptake continue to be concurrently measured. Specifically, participants will step up and down on an aerobic step at 88 beats per minute, dribble a basketball, and perform jumping jacks at 126 beats per minute (63 jumping jacks per minute). Each activity will last for 5 minutes and a 2-minute rest will occur between each activity.

Free-Living, At-Home Monitoring

* Each participant's free-living physical activity will be monitored for 7 whole consecutive days using an ActiGraph GT9X accelerometer positioned on the waist. Participants will wear the accelerometer for 24 hours a day and be asked to maintain their usual lifestyle.
* Participants will complete a physical activity monitoring log, where they will indicate bedtimes, waketimes, and times when the monitor is removed for bathing, swimming, etc.

Visit 2

* Upon returning their free-living wearable monitor and physical activity log, participants will wear a Polar H10 Heart Rate Monitor and a K5 Portable Metabolic Unit during the second visit.
* Cardiorespiratory fitness will be measured by a VO2Peak test, conducted on a treadmill. Participants will walk at a moderate speed, between 2.5 and 3.5 mph. Data collection will begin following completion of a 3-minute warm-up at 0% incline. During the first minute of this warm up, the participant will walk at 1.5 mph. There will be a 1-minute transition period where the treadmill speed will increase to a fast walking speed (2.5-3.5 mph), and another minute will be spent at this speed. The speed determined at the transition period will stay the same for the duration of the test. The treadmill incline will then increase from a 0% incline to a 2% incline. The incline will increase by 2% every two minutes for the first 2 intervals, and then by 1% every minute thereafter.
* Although highly unlikely, if someone continues past the 18% grade, the speed will be increased by 0.2 mph every minute until the test is terminated.
* Rate of perceived exertion will be measured during the last 15 seconds of each testing bout. Gas exchange and heart rate will be monitored continuously.

Visit 3

* Short distance walk

  * Participants will perform a series of self-paced (normal, slow, fast) walks over an electronic, pressure sensitive walkway.
  * Cadence will be determined using data from the pressure sensitive walkway and will inform the speeds used in the following overground walk protocol.
* Overground walk

  * Participants will be fitted with multiple wearable devices (e.g., Fitbit, Apple Watch) to measure/monitor physical activity throughout the testing session.
  * Participants will also wear headphones and be instructed to match their step timing to the tempo they hear in the headphones.
  * After conducting a practice lap, participants will perform five 5-minute overground walks around two, 84 foot by 50 foot basketball courts, each at a different walking speed and to a different tempo played through the headphones. The first three will be at a tempo corresponding to the self-selected slow, normal, and fast walking cadences determined during the short distance walk, respectively. The fourth and fifth tempos will correspond to moderate and vigorous intensity physical activity cadences identified from our previous CADENCE-Kids pilot study (1; NCT01989104). Participants unable to match their steps to the tempo during the practice lap will perform additional laps with the guidance of a pacer. The pacer will walk directly behind participants and support the step timing by verbalizing 'LEFT/RIGHT' at the appropriate timing.
  * Participants will walk over the pressure sensitive walkway every time they complete a lap around the courts, and may walk over the pressure sensitive walkway more than once during each of the 5 bouts.
  * A lab member will manually count total steps for each bout via hand tally. Video recording of participants' lower body movements will be taken to provide redundant step-counting. Digital data displayed on the screens of the wearable devices will be reported at the end of each bout, and data from these wearables will be downloaded after data collection is complete.

ELIGIBILITY:
Inclusion Criteria:

* Between 6 - 20 years of age on the day of signing the informed consent/assent.
* Able to walk without the need of assistance

Exclusion Criteria:

* Need for assistance with walking including the use of a wheelchair
* Mental illness requiring hospitalization within the past 5 years
* Medical condition or medications that affect(s) changes in heart rate with exercise
* Current pregnancy
* Pacemaker or other implanted medical device including metal joint replacements
* History of cardiovascular disease, stroke, transient ischemic attacks (TIA, mini-stroke), chest pain, unusual shortness of breath during physical activity/exercise, swelling in legs/ankles, or excessive leg pain with exercise.
* History of musculoskeletal problems that cause pain during physical activity which interferes with the ability to walk
* Exercise-induced asthma requiring medications prior to low intensity activities like walking
* Unavailable for the entire duration of the study period

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Cadence (steps per minute) | Over the course of the study period (up to 3 months) across 3 visits plus an at-home free-living protocol per participant (see Protocol/Procedures)
  Cadence (steps per minute) represents an overlooked opportunity to describe the intensity of ambulatory activity.

CONTACTS AND LOCATIONS:
Overall Officials: Catrine Tudor-Locke, PhD, Principal Investigator — University of North Carolina at Charlotte; Laura H Gunn, PhD, Principal Investigator — University of North Carolina at Charlotte
Locations (1):
- University of North Carolina at Charlotte, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified dataset will be published along with open-access manuscripts as a supplemental file and available to anyone accessing the article. Requests for de-identified individual-level data (including descriptors) collected in SKyRoCKeT and used in publications will be considered and made available to qualified researchers, in accordance with the NIH Data Sharing Policy and Final NIH Statement on Sharing Research Data. Data sharing agreements will be necessary for access. The SKyRoCKeT database will be maintained and access ensured by SKyRoCKeT team members at the University of North Carolina at Charlotte.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available upon manuscript publication of the full study cohort.
Access Criteria: Requests for de-identified individual-level data (including descriptors) collected in SKyRoCKeT and used in publications will be considered and made available to qualified researchers within 2 years of publication of the associated paper. Data sharing agreements will be necessary for access.

REFERENCES:
- [Background] Tudor-Locke C, Schuna JM Jr, Han H, Aguiar EJ, Larrivee S, Hsia DS, Ducharme SW, Barreira TV, Johnson WD. Cadence (steps/min) and intensity during ambulation in 6-20 year olds: the CADENCE-kids study. Int J Behav Nutr Phys Act. 2018 Feb 26;15(1):20. doi: 10.1186/s12966-018-0651-y. PMID 29482554